CLINICAL TRIAL: NCT01927510
Title: Pilot Randomised Controlled Trial of Early Mobilisation in Critically Ill Patients to Improve Functional Recovery and Quality of Life.
Brief Title: TEAM: A Trial of Early Activity and Mobility in ICU
Acronym: TEAM-RCT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Australian and New Zealand Intensive Care Society Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCT01927510
Record Dates: First submitted 2013-08-15; First posted 2013-08-22 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2015-06

CONDITIONS: Critically Ill
Keywords: Early mobilization, rehabilitation, intensive care
MeSH Terms: conditions — Critical Illness | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early mobilisation (Experimental): intervention of early mobilisation
  Interventions: Behavioral: Early mobilisation
- Control (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Early mobilisation
  Other Names: Rehabilitation
  Arms: early mobilisation

SUMMARY:
Patients in the intensive care unit (ICU) traditionally receive bed rest as part of their care. They develop muscle weaknesses even after only a few days of mechanical ventilation that may prolong their time in ICU and in hospital, delay functional recovery and delay their return home and to work. Weakness may be avoided with simple strategies of early exercise in ICU. This pilot study aims to test the hypothesis that early mobilisation may improve functional recovery in this patient group and gather pilot data to support a larger randomised trial across Australia and New Zealand.

DETAILED DESCRIPTION:
Patients who are admitted and treated in the intensive care unit (ICU) generally have potentially reversible critical illness. While many patients survive, substantial proportions of patients fail to recover completely and do not return to their pre-morbid level of health. Critically ill patients receive mechanical ventilation, as a lifesaving intervention, but this is routinely managed with deep sedation and immobility, which results in prolonged periods of bed rest. Severe muscle weakness, termed ICUAW, is common and associated with prolonged duration of mechanical ventilation and hospital stay in the ICU, as well as poor recovery of physical function. Early mobilisation, exercising patients while they are still receiving mechanical ventilation, has been proposed as a candidate intervention to prevent ICU acquired weakness (ICUAW). Observational studies indicate that early mobilisation is not used routinely in critically ill patients in Australia and New Zealand. TEAM is a pilot RCT designed to obtain data to assist in the planning of an adequately powered RCT that will test the hypothesis that early mobilisation of critically ill patients improves one or more functional outcomes, quality of survival, and proportion of patients who survive.

ELIGIBILITY:
Inclusion Criteria:

* Adults > or + to 18 years old admitted to the ICU
* Invasively ventilated and expected to be ventilated the day after tomorrow
* Written informed consent from person responsible/ net of kin (or consent as per individual HREC if delayed or telephone consent is acceptable)

Exclusion Criteria:

1. INSTABILITY A. Cardiovascular

   * Unresolved rhythm disturbance with any bradycardia requiring pharmacological support
   * Any tachycardia with ventricular rate > 150 beats/min
   * Lactacte > 4.0 due to inadequate tissue perfusion
   * Any external mechanical cardiovascular support (eg. VA ECMO or intra-aortic balloon pump)
   * Norad > 0.2mcg/kg/min (or unit equivalent) or any dose of norad between 0.1 and 0.2mcg/kg/min with more than a 25% increase in last 6 hours
   * Cardiac index < 2.0L/min/m^2

   B. Respiratory
   * FiO2 > 0.6
   * PEEP > 15
   * Requirement for hypoxaemic rescue interventions eg. NO, prone, ECMO, prostacyclin, HFOV
   * RR > 45
2. Proven or suspected actue brain injury such as stroke, sub-arachnoid haemorrhage, encephalitis, or moderate to severe traumatic brain injury
3. Proven or suspected actue spinal cord injury
4. Proven or suspected Guillain-Barre Syndrome
5. Second or subsequent ICU admission during a single hospital admission
6. Unable to follow simple verbal commands in English
7. Death inevitable and imminent
8. Inability to walk without assistance of another person prior to onset of acute illness necessitating ICU admission
9. Cognitive impairment prior to current acute illness
10. Agitation which int he opinion of the treating clinician precludes safe implementation of EGDM
11. Written rest in bed orders due to documented injury or process the precludes mobilisation such as suspected or proven instability of spine or pelvis
12. In the opinion of the treating clinician it is unsafe to commence EGDM
13. Has met all the inclusion criteria with no concomitant exclusion criteria for a period of more than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Highest daily level of activity measured using the ICU mobillity scale | Duration of ICU stay (an average of 10 days)
  ICU Mobility Scale - ranges from 0 (Nothing/Lying in Bed) to 10 (Walking Independently without a Gait Aid)
Total Duration of Active Mobilisation | Radomisation to removal of invasive ventilation (an average of 7 days)
Mean (or Median) Daily Duration of Active Mobilisation | Randomisation to removal of invasive ventilation (daily for an average of 7 days)
  Measured in minutes, any mobilisation activity where the patient can use their own muscle force to assist the movement.
Total Duration of Active Mobilisation | Randomisation to ICU discharge, an average of 10 days
  Pt will be free of Mechanical Ventilation, Vasopressors and Continuous Renal Replacement Therapy for 24 Hours
Mean (or Median) Daily Duration of Active Mobilisation | Randomisation to Time of Final Listing for Ward Discharge, an average of 10 days
  Pt will be free of Mechanical Ventilation, Vasopressors and Continuous Renal Replacement Therapy for 24 Hours (approximately 10 days)
Proportion of Patients achieving each Category of Highest Level of Mobilisation on Each Day | Randomisation to Extubation, an average of 7 days
  Measured using the ICU mobility scale (0-10)

SECONDARY OUTCOMES:
Physical Function | At 6 months from randomisation
  Highest level of activity, measured using the IADL
Recruitment Rates | Entirety of Study
Staff Utilisation Costs | ICU admission (approximately 10 days)
  Number of staff required for mobilisation, minutes spent with the patient on active mobilisation activities, and type of staff such as assistant, physiotherapist or nurse, and specific equipment used during mobilisation ie: tilt table/standing frame.
Ventilator and IC free days at Day 28 | Randomisation to Day 28
  Intensive care free defined as ward ready; free of inotropes, RRT and mechanical ventilation for 24 hours and remaining free of these supports until the time of actual ICU discharge
Health related quality of life | 6 Months after ICU admission
  EQ5D measured using a trained, blinded assessor via telephone interview
Return to previous work level | At 6 months from randomisation
  Has the participant returned to the work level prior to critical illness?

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Hodgson, PhD, Study Chair — Australian and New Zealand Intensive Care Research Centre
Locations (5):
- Australia (3):
  - The Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- New Zealand (2):
  - Auckland CIty Hospital CVICU, Grafton, Auckland
  - Wellington Hospital, Newtown, Wellington Region

REFERENCES:
- [Background] Hodgson CL, Bailey M, Bellomo R, Berney S, Buhr H, Denehy L, Gabbe B, Harrold M, Higgins A, Iwashyna TJ, Papworth R, Parke R, Patman S, Presneill J, Saxena M, Skinner E, Tipping C, Young P, Webb S; Trial of Early Activity and Mobilization Study Investigators. A Binational Multicenter Pilot Feasibility Randomized Controlled Trial of Early Goal-Directed Mobilization in the ICU. Crit Care Med. 2016 Jun;44(6):1145-52. doi: 10.1097/CCM.0000000000001643. PMID 26968024